CLINICAL TRIAL: NCT05983679
Title: Prevalence of Sexually Transmitted Infections (STIs) and Co-infections in the General Population
Brief Title: Prevalence of Sexually Transmitted Infections (STIs) and Coinfections in the General Population
Acronym: PREMINF
Status: Not yet recruiting | Type: Observational
Sponsor: CerbaXpert (Other)
Responsible Party: Sponsor
Other Study IDs: PREMINF
Record Dates: First submitted 2023-06-22; First posted 2023-08-09 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults
  Interventions: Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: Blood sample — Blood sample

SUMMARY:
Prevalence of Sexually Transmitted Infections (STIs) and co-infections in the general population

ELIGIBILITY:
Inclusion Criteria:

* Subject, male or female, 18 years of age or older
* Subject capable of understanding the purpose of the research having given their free and informed written consent
* Subject presenting to the laboratory for a biological examination
* Affiliated subject or beneficiary of a social security scheme

Exclusion Criteria:

- Protected subject: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A cohort of 9,000 participants meeting all the inclusion criteria will be recruited. A participant identification list will be created and maintained at clinical investigation sites, linking the participant's personal data to the code assigned in the research. The identification list of participants will be kept on the research site in paper or digital format classified in the investigator binder.
Sampling Method: Probability Sample
Enrollment: 9000 (Estimated)
Dates: Start 2024-12-04 (Estimated); Primary Completion 2025-09-04 (Estimated); Study Completion 2026-09-04 (Estimated)

PRIMARY OUTCOMES:
The prevalence of each STI will be assessed by the participant's positive or negative status for each pathogen, determined by the following screening tests: | 3 years
  HIV testing is based on finding antibodies to HIV-1 and HIV-2 and P24 antigen of the virus;
  * Hepatitis B screening is based on HBsAg (hepatitis B surface antigen) research;
  * Herpes screening is based on testing for antibodies to Herpes Simplex virus (HSV-1 and HSV-2);
  * Papilloma virus screening is based on the HPV-HR test from a smear on the cervix;
  * Chlamydia screening is based on a nucleic acid amplification (NAAT) test;
  * Gonorrhea screening is based on the identification of the bacteria on a urine sample or secretions from the vagina or cervix;
  * Screening for trichomoniasis is based on a molecular diagnosis that involves identifying the parasite's DNA from a genital or urinary sample;
  * The detection of syphilis is based on antibody research.

IPD SHARING:
Plan to Share IPD: No